CLINICAL TRIAL: NCT04874662
Title: Efficacy and Safety of a Mix of Nicotinamide (NAM) and Pyridoxine (vitamin B6) on Muscle Regeneration: a Randomized, Double-blind, Placebo-controlled Study ("Satellite-01 Study").
Brief Title: Nicotinamide (NAM) and Pyridoxine (vitamin B6) on Muscle Regeneration ("Satellite-01 Study").
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20.07.CLI
Record Dates: First submitted 2021-05-04; First posted 2021-05-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Muscle Injury

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational NAM/B6 (Active Comparator): 2 VCaps® capsules daily (commercial vegetarian capsules made of Hydroxy Propyl Methyl Cellulose, a polymer of cellulose)
  Dosage per capsule: 357mg of nicotinamide, 9.5mg of pyridoxine and 195mg of microcrystalline cellulose
  Form:The VCaps® Size 00 will be used. They have a volume of 0.95 ml for 23.3 mm length and a diameter of 8.51 mm head / 8.16 mm body.daily of NAM/B6
  Frequency and duration: 2 capsules daily for 9 days
  Interventions: Dietary Supplement: NAM/B6
- Placebo control group (Placebo Comparator): 2 capsules daily of microcrystalline cellulose excipient (337mg per capsule)
  Frequency and duration: 2 capsules daily for 9 days
  Interventions: Dietary Supplement: NAM/B6

INTERVENTIONS:
Dietary Supplement: NAM/B6 — Single daily dose administration will take place from Day 0 (V1) to Day 8 (V4) around 8 am after an overnight fast from the subsequent evening at 9 pm.

SUMMARY:
Assessment of safety and efficacy of NAM/B6 oral administration on the amplification and commitment of satellite cells after a muscle injury

DETAILED DESCRIPTION:
NAM/B6 oral administration after a muscle injury ("Satellite-01 study"): Effect on satellite cells as measured by immunofluorescence (Pax7 and myogenin antibodies to detect amplifying and committed satellite cells, respectively) on sections of muscle biopsies from the stimulated leg (leg 2) by muscle biopsies, comparing the study intervention (NAM/B6) to the control intervention (placebo)

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥18 ≤ 50 years;
2. Subjects must be in good general health, as determined by the investigator or delegate, based on a comprehensive medical evaluation at screening including detailed medical history, full physical examination, blood pressure and heart rate measurements, 12-lead electrocardiogram (ECG) and clinical laboratory tests;
3. Body mass index (BMI) between18.5 and 24.9 kg/m2;
4. Normal dietary habits;
5. Willing to adhere to the prohibitions and restrictions specified in the protocol;
6. Must understand the nature of the study and be capable of giving written informed consent and be willing to report for the scheduled study visits and communicate to study personnel about adverse events and concomitant medication use.

Exclusion Criteria:

1. Subjects presenting with the following blood pressure (BP) and heart rate (HR) values at the screening visit after 10 minutes in supine position:

   1. 95 mmHg ≤ systolic blood pressure (SBP) ≤ 140 mmHg,
   2. 50 mmHg ≤ diastolic blood pressure (DBP) ≤ 95 mmHg,
   3. 50 bpm < HR < 80 bpm,
   4. Or any other out of expected range values considered clinically significant by the investigator;
2. Screening visit 12-lead ECG values which are:

   1. 120 < PR segment < 220 ms,
   2. QRS complex < 120 ms,
   3. QTcf < 430 ms,
   4. Sign of any trouble of sinusal automatism,
   5. Or any other ECG finding considered clinically significant by the investigator;
3. Have any clinically significant abnormalities in serum chemistry, hematology, or urinalysis at screening as judged by the investigator or delegate;
4. Active smokers;
5. Vegetarians or vegans;
6. Performed structured exercises within 3 months prior to participation in the study;
7. History or current use of anabolic steroids and/or growth hormone;
8. Use of corticosteroids within 3 months prior to participation in the study;
9. Current use of anticoagulant or anti-aggreging agents;
10. History or current use since 2 weeks before inclusion of any of the prohibited medications as detailed in Section 6.6.2;
11. History or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, musculoskeletal, psychiatric, systemic or infectious disease;
12. History or current use of drugs or alcohol (alcohol consumption > 40 grams/day);
13. Known intolerance to foods containing the ingredients under investigation;
14. Knee pain that prevents application of the electrical muscle stimulation protocol;
15. Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
16. Subjects under administrative or legal supervision;
17. Have participated in a clinical study in the last 3 months and received compensation beyond a certain approved and predefined limit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
immunofluorescence measurement | 9 days
  Number of satellite cells as measured by immunofluorescence (Pax7 and myogenin antibodies to detect amplifying and committed satellite cells, respectively) on sections of muscle biopsies from the stimulated leg (leg 2) at day 4 and day 8 (muscle biopsies: MB3 and MB5), comparing the study intervention (NAM/B6) to the control intervention (placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, Prof, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Bisepjerg-Frederiksbjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No